CLINICAL TRIAL: NCT00004073
Title: Phase II Study of Suramin and Concurrent Radiation Therapy in Newly Diagnosed Glioblastoma Multiforme
Brief Title: Suramin Plus Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTT-9808 CDR0000067281; U01CA062475 (NIH); P30CA006973 (NIH); NABTT-9808; JHOC-NABTT-9808
Record Dates: First submitted 1999-12-10; First posted 2004-05-20 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Suramin; Radiotherapy

INTERVENTIONS:
Drug: suramin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Suramin may stop the growth of glioblastoma multiforme by stopping blood flow to the tumor. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining suramin with radiation therapy may be a more effective treatment for glioblastoma multiforme.

PURPOSE: Phase II trial to study the effectiveness of suramin plus radiation therapy in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity of suramin administered prior to and concurrent with radiotherapy in patients with newly diagnosed high grade glioblastoma multiforme. II. Evaluate this regimen in terms of survival in this patient population.

OUTLINE: Patients receive suramin IV over 2 hours for initial dose and over 1 hour for subsequent doses daily for 5 days on week 1. Patients receive concurrent radiotherapy daily with suramin IV over 1 hour twice weekly on weeks 2-7. Patients with stable or responsive disease receive a second course of suramin twice weekly on weeks 20-24. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months until disease progression or start of new therapy and then monthly for survival.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study over 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed supratentorial glioblastoma multiforme No prior intracranial or intratumoral hemorrhage

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Greater than 2 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL No history of a bleeding disorder that would interfere with protocol therapy Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases no greater than 4 times upper limit of normal Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: No suspected disseminated intravascular coagulation No history of venous thrombosis requiring coumadin Other: No serious concurrent infection or other medical illness that would prevent compliance No other malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy or biologic agents (e.g., immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, lymphokine activated killer cells, tumor infiltrating lymphocytes, or gene therapy) for brain tumor Chemotherapy: No prior chemotherapy for brain tumor Endocrine therapy: No prior hormonal therapy for brain tumor Prior glucocorticoids allowed Maintenance 5 day stable corticosteroid regimen required postsurgery Radiotherapy: No prior radiotherapy for brain tumor Surgery: Prior surgery for brain tumor allowed if recovered from the immediate post operative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 1999-12; Primary Completion 2003-05 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Laterra, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (9):
- United States (9):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Laterra JJ, Grossman SA, Carson KA, Lesser GJ, Hochberg FH, Gilbert MR; NABTT CNS Consortium study. Suramin and radiotherapy in newly diagnosed glioblastoma: phase 2 NABTT CNS Consortium study. Neuro Oncol. 2004 Jan;6(1):15-20. doi: 10.1215/S1152851703000127. PMID 14769135